CLINICAL TRIAL: NCT01839929
Title: A Multicenter, Open-label, Single-arm, Non-inferiority Study to Assess the Safety and Efficacy of a Tacrolimus Modified Release, ADVAGRAF® in Stable Kidney Transplant Patients Converted From a PROGRAF® Based Immunosuppressive Regimen
Brief Title: A Study to Assess the Safety and Efficacy of ADVAGRAF (Tacrolimus Modified Release Formulation) in Kidney Transplant Patients Who Were Treated With PROGRAF
Acronym: PeACE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADV-KT-02
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Kidney Transplantation
Keywords: tacrolimus; immunosuppressant; FK506
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prograf/Advagraf (Experimental): conversion from Prograf to Advagraf
  Interventions: Drug: Prograf; Drug: Advagraf

INTERVENTIONS:
Drug: Prograf — oral
  Other Names: FK506; tacrolimus
Drug: Advagraf — oral
  Other Names: FK506E; tacrolimus modified release formulation

SUMMARY:
The purpose of this study is to evaluate the efficacy of tacrolimus modified release formulation Advagraf® after conversion from Prograf® in stable kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients received a kidney transplant at least 12 months ago prior to enrollment.
2. Patients have taken unchanged dosage of Prograf® and remained stable serum level of tacrolimus at least for 12 weeks prior to enrollment.
3. Patients have kept in unchanged immunosuppressive therapy (combination therapy) at least for 12 weeks prior to enrollment.
4. Female patients of childbearing potential must have a negative urine or serum pregnancy test prior to enrollment, and agreed to the deliberate prevention of conception during the trial.
5. Patients are considered clinically stable by observer's judgment.
6. Patients must understand the purpose and risk of participating the trial and signed on the written consent.

Exclusion Criteria:

1. Patients have previously received an organ transplant other than a kidney.
2. Patients have had acute transplant rejection within 12 weeks, or acute transplant rejection requiring antilymphocyte therapy within 24 weeks prior to enrollment.
3. Patients newly diagnosed malignant tumors after organ transplant but the patients treated completely with basal or squamous cell carcinoma of the skin are excepted.
4. Patients have a known hypersensitivity to Prograf® or tacrolimus.
5. Patients whose medical condition are able to interfere with the study objectives.
6. Patients who are at the risk of drug abuse or mental disorders or communicate difficulties with the observer.
7. Patients have been participated in another clinical trial, or treated with drugs of clinical trial within 28 days prior to enrollment.
8. Patients have been taken prohibited combination agents within 28 days prior to enrollment.
9. Patients are pregnant or lactating.
10. Patient are HIV-positive.
11. Patients are not able to keep the scheduled visit.
12. Patients whose GFR (MDRD) is in the level of <30 mL/min.
13. Patients who are at the condition of 'Creeping creatinine (defined by 20% increase within 6 months prior to enrollment)
14. Patients whose SGPT/AST and/or SGOT/ALT levels have been elevated greater than 2 times the upper value of the normal range.
15. Patients have FSGS or MPGN Type II as underlying diseases.
16. Patients are with cirrhosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2010-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change in glomerular filtration rate (GFR) at Week 24 from baseline | Baseline and Week-24

SECONDARY OUTCOMES:
Change in Blood Pressure (BP) at Week 24 from baseline | Baseline and Week-24
Change in HbA1c at Week 24 from baseline | Baseline and Week-24
Change in tacrolimus blood trough level at Week 24 from baseline | Baseline and Week-24
Safety assessed by the incidence of adverse events, physical exam., vital signs and labo tests | For 24 weeks
Overall frequency of acute rejection | For 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Korea, Inc.
Locations (4):
- South Korea (4):
  - Busan
  - Daegu
  - Daejeon
  - Seoul